CLINICAL TRIAL: NCT05602324
Title: Nutritional Supplement for Patients With Severe Infection
Acronym: NUWISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, john boyd, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-00109
Record Dates: First submitted 2022-10-26; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Severe Infection
Keywords: dyslipidemia
MeSH Terms: conditions — Infections; Dyslipidemias | interventions — lauric acid; Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lauric Acid and Berberine (Experimental): Participants in this arm of the trial will receive 15 ml lauric acid and 1000 mg berberine daily (via feed tube) for the duration of time that they are receiving enteral feeding, up to a maximum time of 14 days
  Interventions: Dietary Supplement: Lauric Acid and Berberine
- No-intervention (No Intervention): participants in this arm will receive no additional intervention, beyond standard of care

INTERVENTIONS:
Dietary Supplement: Lauric Acid and Berberine — intervention (15 ml lauric acid + 1000 mg berberine) will be provided daily to participants in this arm for the duration of time that they receive enteral nutrition for a period of 14 days maximum
  Arms: Lauric Acid and Berberine

SUMMARY:
This is a randomized trial testing a supplement that has been approved by Health Canada to support healthy cholesterol levels (i.e. high density lipoprotein (HDL) cholesterol). This trial is proposing to use this approved supplement to determine whether it is able to raise HDL cholesterol in patients treated in the intensive care unit (ICU) with severe infection who have detrimentally low levels of HDL cholesterol. Patients who present to the ICU with severe infection will be approached for consent. If they choose to participate, patients will be given usual care or a 150mL daily nutritional supplement containing lauric acid (15 ml) and Berberine (1000 mg) daily for 14 days. Participants will be followed during their stay in the ICU and will receive follow up phone calls at Day 28 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Sepsis
* plasma high density lipoprotein levels less than 1 mM
* receiving enteral nutrition

Exclusion Criteria:

• known pregnancy/intending to get pregnant within 28 days of enrollment in study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Plasma HDL | 14 days
  Maximum Plasma Concentration [Cmax] HDL (mmol)

SECONDARY OUTCOMES:
WBC | 14 days
  Absolute count (cells per microliter)
Cytokines | 14 days
  Maximum Plasma Concentration [Cmax] plasma IL-6, IL-8, IL-10
28-day survival | 28 days
  28-day survival

CONTACTS AND LOCATIONS:
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
we are in the process of developing a plan to share data from this study